CLINICAL TRIAL: NCT03090854
Title: Cholinergic Markers as Predictive Tools of Therapeutic Response in Alzheimer's Disease (CHOLINE)
Brief Title: Cholinergic Markers Alzheimer's Disease
Acronym: CHOLINE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K160402; 2016-AO1639-42 (Other: IDRCB)
Record Dates: First submitted 2017-02-20; First posted 2017-03-27 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Cognition; Cholinergic target
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alzheimer disease patients
  Interventions: Diagnostic Test: ADASCog

INTERVENTIONS:
Diagnostic Test: ADASCog — Neuropsychological test

SUMMARY:
Several previous studies have assessed acetylcholine (Ach) and acetylcholinesterase activity (AchE-a) levels in Alzheimer's disease (AD) pathophysiology. The cerebrospinal fluid (CSF) Ach level was significantly decreased in AD patients, and correlated positively with dementia score and MMSE (1, 2). Two studies have demonstrated positive correlations between CSF AchE-a and CSF Tau, phosphorylated-Tau (P-Tau) and AB 1-42 peptide (3,4). ChEIs (cholinesterase inhibitors) have been approved for the treatment of AD but only 20 to 30 % of patients are responders (5). Any consistent data allow the clinician to predict the response to the treatment. The link between basal cholinergic status and ChEIs efficiency has never been done. Even if, there is a wild research in AD treatment, ChEIs or treatment acting on the Ach pathways will remain a long time valuable treatment particularly in moderate AD in which disease modifying therapies did not show any efficiency.

The investigators's objective is to prospectively explore the predicting value of CSF Ach and AchE-a levels on ChEIs response in AD patients.

DETAILED DESCRIPTION:
Strategy: Within the framework of the usual management, the investigators propose the protocol to patients who had an assay of the CSF biomarkers with a CSF AD biological profile before the introduction of an IChEs and having accepted Their CSF will stocked in our biobank. Patients will only have additional neuropsychological assessments. The rest of the care comes under the current care.

The quantification of ACh in the CSF will be performed in tandem mass spectrometry after separation by liquid chromatography (LC-MS / MS). AChE activity will be determined by colorimetric determination.

The investigators's objective is to prospectively explore the predicting value of CSF Ach and AchE-a levels on ChEIs response in AD patients.

The evaluation criteria will be

* Difference of the mean value of the ACh level and AChE activity in the CSF between the responder and non-respondier groups of patients.
* "Responder" patients are defined by an improvement of at least 4 points on the ADAS-Cog (cognitive part) ADAS-Cog after 6 months of treatment.
* "Non-responders" are defined as aggravation, lack of improvement or improvement <4 points on the ADAS-Cog scale.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria :

* Male or Female aged ≥ 50 years
* Patients with a biological profile of CSF biomarkers in favor of Alzheimer's disease
* Alzheimer's disease diagnosed according to McKahnn 2011 criteria [1] at mild to moderate stage Clinical Dementia Rating (CDR) ≤2
* Indication to treatment with inhibitor of acetycholinesterase
* Patients benefiting from national health coverage
* Patients not subject to legal protection
* Fluent in French language

Exclusion criteria :

* No indication or contraindication to PL
* Contraindications to IChEs
* Patient included in other anti-Alzheimer drug clinical trial
* Clinical Dementia Rating CDR> 2
* Another cause of neurocognitive decline
* Serious psychiatric disorders
* Other serious life-threatening conditions

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mild to moderate Alzheimer disease 's patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Neuropsychological test (ADASCog) | between baseline and month 6
  "Responder" patients are defined by an improvement of at least 4 points on the ADAS-Cog (cognitive part) ADAS-Cog after 6 months of treatment. "Non-responders" are defined as aggravation, lack of improvement or improvement <4 points on the ADAS-Cog scale

SECONDARY OUTCOMES:
Rate of responder AD in this cohort included according to the new AD criteria and comparison of the current rate with the previous rate published using former AD criteria | month 6
  Alzheimer disease (AD)
Difference of CSF Ach AND AChE activity between responder and non responder groups | month 6
  biological test
Statistical evaluation of the link between CSF Ach, AChE activity, total and phosphorylated Tau, Aß40 and Aß42. | month 6
  biological test

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Mémoire de Ressources et de Recherche Paris Nord, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided